CLINICAL TRIAL: NCT02240186
Title: Comparative Effectiveness Between Microprocessor Knees and Non-Microprocessor Knees
Acronym: MPK-AOPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: American Orthotic and Prosthetic Association (Other)
Responsible Party: Principal Investigator, Kenton R. Kaufman, Ph.D., Professor of Biomedical Engineering, College of Medicine, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-002930; Foundation (Other Grant/Funding Number: American Orthotic and Prosthetic Association)
Record Dates: First submitted 2014-09-08; First posted 2014-09-15 (Estimated); Results first posted 2018-12-12 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Lower Limb Amputation Above Knee (Injury)
Keywords: Microprocessor-controlled knee; prosthesis; amputation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Prosthetic knee joints (Experimental): Each subject will be tested using their current Non-Microprocessor Knee (NMPK) , fit and tested with a Microprocessor Knee (MPK), and then tested again with their NMPK, e.g. A-B-A design.
  Interventions: Device: Microprocessor Knee (MPK); Device: Non-Microprocessor Knee (NMPK)

INTERVENTIONS:
Device: Microprocessor Knee (MPK) — MPKs are prosthetic knees that use a microprocessor to control the prosthetic knee mechanism and adjust knee stiffness.
Device: Non-Microprocessor Knee (NMPK) — A NMPK is a mechanical knee with either hydraulic or pneumatic controls.

SUMMARY:
This study will assess if the functional performance and musculoskeletal outcome of transfemoral amputees are improved after receiving a Microprocessor Knee (MPK) compared to a Non-Microprocessor Knees (NMPK).

DETAILED DESCRIPTION:
The study design is a reversal design whereby only the prosthetic knee joint will be changed. Each subject will be tested using their current NMPK, fit and tested with a MPK, and then tested again with their NMPK. MPK prostheses from all manufacturers will be considered appropriate for testing. Each MPK to be used in this study is FDA approved. The foot will be in the L5981 class, e.g. flex foot or equivalent. The same socket, suspension, and foot will be used throughout the study in order to eliminate these confounding variables. All prosthesis fittings will be performed by the subject's own certified prosthetist according to manufacturers' fitting guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral amputee
* Medicare Functional Classification Level K2 or K3
* Currently using NMPK prosthesis
* No current residual limb problems, such as skin breakdown
* Able to ambulate without a gait aid

Exclusion Criteria:

* Previous stroke or other neuromuscular complications currently affecting gait
* Currently undergoing dialysis treatments
* Amputation of the contralateral limb
* Poor fit of current NMPK prosthesis

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-06 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenton R Kaufman, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Result] Kaufman KR, Bernhardt KA, Symms K. Functional assessment and satisfaction of transfemoral amputees with low mobility (FASTK2): A clinical trial of microprocessor-controlled vs. non-microprocessor-controlled knees. Clin Biomech (Bristol). 2018 Oct;58:116-122. doi: 10.1016/j.clinbiomech.2018.07.012. Epub 2018 Jul 19. PMID 30077128

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prosthetic Knee Joints
Started | 50
Completed | 23
Not Completed | 27

BASELINE CHARACTERISTICS:
Arm/Group | Prosthetic Knee Joints
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 28
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Daily Activity Measured With Triaxial Accelerometers
Description: Measurements will be obtained three times using activity monitors attached to waist, and bilaterally to the ankle and thigh for a period of 4 consecutive days, including 2 weekdays and 2 weekend days. Primary outcome will be the difference in activity level between the NMPK and MPK measurements.
Time Frame: Baseline (tested on subjects' current NMPK), 10 weeks (after 10 weeks acclimation time to the study MPK) , 4 weeks (subjects placed back on NMPK and tested after 4 weeks re-acclimation time)
Population: Activity measurement data were available for analysis on 46 baseline participants, 31 MPK participants, and 18 NMPK participants.
Measure: Mean (Standard Deviation); unit: % of Day
Arm/Group | Prosthetic Knee Joints
Number analyzed (Participants) | 46
% of Day
  Baseline | 15.64 (8362)
  MPK: number analyzed (Participants) | 31
  MPK | 19.68 (11.88)
  NMPK: number analyzed (Participants) | 18
  NMPK | 18.23 (10.54)
Statistical Analysis 1: Comparison: Prosthetic Knee Joints; Test type: Superiority; p = 0.01, ANOVA

2. Primary Outcome: Falls as Assessed by the Prosthesis Evaluation Questionnaire Addendum (PEQ-A)
Description: The Prosthesis Evaluation Questionnaire (PEQ) addendum (PEQ-A) is a self-administered questionnaire to quantify balance confidence, concentration, stumbles, and falls. The outcome will be difference in falls per month between the Non-Microprocessor Knee (NPMK) and MPK measurements. The number of falls was recorded as the sum of items #5 and #7 in the PEQ-A.
Time Frame: as for outcome 1
Population: Data for falls were available for analysis on 46 baseline participants, 30 MPK participants, and 17 NMPK participants.
Measure: Median (Inter-Quartile Range); unit: Falls per month
Arm/Group | Prosthetic Knee Joints
Number analyzed (Participants) | 46
Falls per month
  Baseline | 2.0 [0.0 to 6.0]
  MPK: number analyzed (Participants) | 30
  MPK | 0.0 [0.0 to 3.25]
  NMPK: number analyzed (Participants) | 17
  NMPK | 3.0 [0.0 to 3.0]
Statistical Analysis 1: Comparison: Prosthetic Knee Joints; Test type: Superiority; p = 0.01, ANOVA

3. Secondary Outcome: Patient Satisfaction as Assessed by the Prosthesis Evaluation Questionnaire (PEQ)
Description: The condition-specific Prosthesis Evaluation Questionnaire (PEQ) was used to quantify patient satisfaction with each prosthesis. The outcome was a difference in PEQ scores between the NPMK and MPK measurements.
  The PEQ is a self-administered questionnaire composed of nine validated scales (ambulation, appearance, frustration, perceived response, residual limb health, social burden, sounds, utility, well being). Scores range from 0 to 100 for each sub-scale. Higher scores indicated a higher functioning prosthesis/quality of life.
Time Frame: as for outcome 1
Population: Not all participants completed all the scales in the questionnaire.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Prosthetic Knee Joints - NMPK Baseline; Prosthetic Knee Joint - MPK; Prosthetic Knee Joint - NMPK: Each subject will be tested using their current Non-Microprocessor Knee (NMPK) , fit and tested with a Microprocessor Knee (MPK), and then tested again with their NMPK, e.g. A-B-A design.
  Microprocessor Knee (MPK): MPKs are prosthetic knees that use a microprocessor to control the prosthetic knee mechanism and adjust knee stiffness.
  Non-Microprocessor Knee (NMPK): A NMPK is a mechanical knee with either hydraulic or pneumatic controls.
Arm/Group | Prosthetic Knee Joints - NMPK Baseline | Prosthetic Knee Joint - MPK | Prosthetic Knee Joint - NMPK
Number analyzed (Participants) | 48 | 33 | 23
Score on a scale
  Ambulation: number analyzed (Participants) | 46 | 32 | 20
  Ambulation | 39.07 (17.14) | 49.58 (24.61) | 45.31 (20.94)
  Appearance: number analyzed (Participants) | 47 | 31 | 20
  Appearance | 64.55 (18.81) | 74.43 (20.64) | 62.80 (19.37)
  Frustration: number analyzed (Participants) | 46 | 32 | 19
  Frustration | 51.48 (29.44) | 66.28 (28.67) | 56.29 (28.83)
  Perceived Response: number analyzed (Participants) | 40 | 28 | 17
  Perceived Response | 85.23 (12.29) | 89.28 (12.88) | 90.00 (9.91)
  Residual Limb Health: number analyzed (Participants) | 47 | 32 | 20
  Residual Limb Health | 74.46 (19.95) | 77.08 (15.58) | 76.31 (18.56)
  Social Burden: number analyzed (Participants) | 43 | 29 | 20
  Social Burden | 62.21 (22.75) | 71.71 (23.00) | 66.06 (29.15)
  Sounds: number analyzed (Participants) | 47 | 32 | 20
  Sounds | 76.96 (25.28) | 81.70 (23.22) | 85.13 (16.91)
  Utility: number analyzed (Participants) | 47 | 32 | 20
  Utility | 53.96 (16.48) | 64.09 (21.07) | 52.52 (14.18)
  Well Being: number analyzed (Participants) | 47 | 31 | 20
  Well Being | 53.47 (21.81) | 62.00 (22.18) | 61.10 (20.28)
Statistical Analysis 1: Comparison: Prosthetic Knee Joints - NMPK Baseline vs Prosthetic Knee Joint - MPK; Test type: Superiority; p = 0.01, ANOVA

ADVERSE EVENTS:
Time Frame: Acclimation period through assessment after reversion to the NMPK, up 6 months.
Arm/Group | Prosthetic Knee Joints
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50
Other Adverse Events (participants affected / at risk) | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-09-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT02240186/Prot_SAP_000.pdf